CLINICAL TRIAL: NCT03920865
Title: An Open-Label, Single-Dose, Parallel-Group, Two-Part Study to Evaluate the Pharmacokinetics and Safety of Risdiplam in Subjects With Mild or Moderate Hepatic Impairment Compared to Subjects With Normal Hepatic Function
Brief Title: A Study to Investigate the Effect of Hepatic Impairment on the Pharmacokinetics and Safety and Tolerability of a Single Oral Dose of Risdiplam Compared to Matched Healthy Participants With Normal Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BP40995
Record Dates: First submitted 2019-04-17; First posted 2019-04-19 (Actual); Results first posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-01

CONDITIONS: Muscular Atrophy, Spinal
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — Risdiplam

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 (Experimental): Participants with mild hepatic impairment and demographically matched healthy participants with normal hepatic function will be enrolled. Participants will receive a single oral dose of 5 mg risdiplam.
  Interventions: Drug: Risdiplam
- Part 2 (Experimental): Participants with moderate hepatic impairment and demographically matched healthy participants with normal hepatic function will be enrolled. Participants will receive a single oral dose of 5 mg risdiplam.
  Interventions: Drug: Risdiplam

INTERVENTIONS:
Drug: Risdiplam — 5 milligram (mg) oral dose administered in fasted state

SUMMARY:
This is a multi-center, open-label, non-randomized, parallel-group, 2-part study to evaluate the effect of hepatic impairment on the PK and safety and tolerability of a single oral dose of risdiplam compared to matched healthy participants with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

All Participants:

* BMI between 18.0 and 36.0 kilograms per square metre (kg/m2), inclusive, and body weight > / = 50 kg
* Females must not be pregnant or lactating and must be of non-childbearing potential
* Male participants (whether surgically sterilized or not) with female partners of childbearing potential must use methods of contraception from Screening until 4 months after their dose of the study drug as detailed in the protocol
* Male participants must not donate sperm from Check-in (Day -1) until 4 months after their dose of the study drug

Participants with Normal Hepatic Function Only:

* Matched to participants with mild or moderate hepatic function in sex, age, BMI, and smoking status
* In good health, as determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, vital sign measurements, and clinical laboratory evaluations

Participants with Hepatic Impairment Only:

* Documented chronic stable liver disease
* Currently on a stable medication regimen, defined as not starting new drug(s) or changing drug dose(s) within 3 months of administration of study drug
* Anemia secondary to hepatic disease will be acceptable, if hemoglobin >/= 9 gram per decilitre (g/dL). Participants must have a platelet count </= 35 000 platelets

Exclusion Criteria:

All Participants

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, constituents or excipients of the study drug, food, or other substance
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered
* Ventricular dysfunction or history of risk factors for Torsades de Pointes
* Evidence of hepatorenal syndrome and estimated creatinine clearance range < 60 millilitre per minute (mL/min) or abnormal sodium and potassium levels
* Clinically significant physical examination abnormality
* History of diabetes mellitus
* Use or intend to use any medications/products known to alter drug absorption, metabolism, or elimination processes, including St. John's Wort
* Positive human immunodeficiency virus (HIV) test
* Participation in a clinical study involving administration of an investigational drug prior to dosing
* Smoke more than 10 cigarettes or use the equivalent tobacco- or nicotine-containing products per day
* Receipt of blood products within 2 months prior to study
* Donation of blood, plasma, or platelets prior to Screening
* Poor peripheral venous access
* Have previously completed or withdrawn from this study or any other study investigating risdiplam, and have previously received the investigational product

Participants with Normal Hepatic Function Only:

* Confirmed supine blood pressure > 150 millimetre of mercury (mmHg) or < 90 mmHg
* Positive test for hepatitis B or C virus
* Clinically significant abnormal laboratory values
* Significant history or clinical manifestation of hepatic disorder
* History or presence of liver disease or liver injury
* Use or intend to use any prescription medications/products within 14 days prior to dosing

  -. Use or intend to use slow-release medications/products considered to still be active within 14 days prior to dosing
* Use or intend to use any non-prescription medications/products within 7 days prior to dosing

Participants with Hepatic Impairment Only:

* Confirmed supine blood pressure > 159 mmHg or < 90 mmHg
* Values outside the normal range for liver function tests that are not consistent with their hepatic condition
* Use of a new medication, or a change in dose, for the treatment, or worsening of, hepatic encephalopathy
* Use of prescription drugs within 14 days of study drug administration
* Recent history of, or the treatment of, esophageal bleeding
* Presence of a portosystemic shunt
* Recent history of paracentesis
* Current functioning organ transplant or are waiting for an organ transplant
* Evidence of severe ascites
* History or current symptoms of hepatic encephalopathy Grade 2 or above

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2020-01-02 (Actual); Study Completion 2020-01-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- United States (3):
  - Clinical Pharmacology of Miami, Inc., Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - American Research Corporation Inc., San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.clinicalstudydatarequest.com). Further details on Roche's criteria for eligible studies are available here (https://clinicalstudydatarequest.com/Study-Sponsors/Study-Sponsors-Roche.aspx). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Groups:
- Mild Hepatic Impairment: All participants received a single dose of 5 mg risdiplam orally as a drinking solution on Day 1 after an overnight fast of at least 8 hours in Part 1 of the study.
- Moderate Hepatic Impairment: All participants received a single dose of 5 mg risdiplam orally as a drinking solution on Day 1 after an overnight fast of at least 8 hours in Part 2 of the study.
- Normal Hepatic Function: All participants received a single dose of 5 mg risdiplam orally as a drinking solution on Day 1 after an overnight fast of at least 8 hours. Two normal function participants were matched as controls for mild hepatic impairment participants in Part 1 only; likewise, two normal function participants were matched to moderate hepatic impairment participants in Part 2 only. Six of the normal function participants were matched to mild hepatic impairment participants in Part 1 and also to moderate impairment participants in Part 2.
Period: Overall Study
Arm/Group | Mild Hepatic Impairment | Moderate Hepatic Impairment | Normal Hepatic Function
Started | 8 | 8 | 10
Completed | 8 | 8 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mild Hepatic Impairment | Moderate Hepatic Impairment | Normal Hepatic Function | Total
Number analyzed (Participants) | 8 | 8 | 10 | 26
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.5 (4.0) | 56.6 (6.3) | 57.3 (6.8) | 58.4 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 5 | 13
  Male | 4 | 4 | 5 | 13
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7 | 14
  Not Hispanic or Latino | 5 | 4 | 3 | 12
Race/Ethnicity, Customized [Number; unit: Participants]
  Black or African American | 2 | 1 | 0 | 3
  White | 6 | 7 | 10 | 23

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity (AUCinf) of Risdiplam and Its Metabolite (M1)
Time Frame: Predose, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264, 312, 336, 360, 408, 456, 504, and 552 hours Postdose
Population: The PK population included all participants who received a dose of risdiplam and had evaluable PK data. A participant was excluded from the PK descriptive statistics and statistical analysis if the participant had an AE of vomiting that occurred at or before 2 times median time to maximum concentration or if they had any major protocol deviation(s) thought to impact PK analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- Risdiplam - Mild Hepatic Impairment; Risdiplam M1 Metabolite - Mild Hepatic Impairment: Participants with mild hepatic impairment received a single dose of 5 mg risdiplam orally as a drinking solution on Day 1 after an overnight fast of at least 8 hours.
- Risdiplam - Normal Hepatic Function; Risdiplam M1 Metabolite - Normal Hepatic Function: Participants with normal hepatic function received a single dose of 5 mg risdiplam orally as a drinking solution on Day 1 after an overnight fast of at least 8 hours.
Arm/Group | Risdiplam - Mild Hepatic Impairment | Risdiplam - Normal Hepatic Function | Risdiplam M1 Metabolite - Mild Hepatic Impairment | Risdiplam M1 Metabolite - Normal Hepatic Function
Number analyzed (Participants) | 8 | 8 | 8 | 8
h*ng/mL | 792 (20.0) | 987 (35.2) | 222 (36.6) | 263 (44.1)
Statistical Analysis 1: Comparison: Risdiplam - Mild Hepatic Impairment vs Risdiplam - Normal Hepatic Function; Test type: Other — Descriptive statistics; Ratio of Geometric Least Squares Means = 0.802, 90% CI 2-sided [0.627 to 1.03]
Statistical Analysis 2: Comparison: Risdiplam M1 Metabolite - Mild Hepatic Impairment vs Risdiplam M1 Metabolite - Normal Hepatic Function; Test type: Other — Descriptive statistics; Ratio of Geometric Least Squares Means = 0.842, 90% CI 2-sided [0.588 to 1.21]

2. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to the Last Measurable Concentration (AUClast) of Risdiplam and M1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Risdiplam - Mild Hepatic Impairment | Risdiplam - Normal Hepatic Function | Risdiplam M1 Metabolite - Mild Hepatic Impairment | Risdiplam M1 Metabolite - Normal Hepatic Function
Number analyzed (Participants) | 8 | 8 | 8 | 8
h*ng/mL | 773 (20.3) | 961 (35.9) | 197 (39.1) | 245 (47.1)

3. Primary Outcome: Part 1: Maximum Observed Plasma Concentration (Cmax) of Risdiplam and M1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Risdiplam - Mild Hepatic Impairment | Risdiplam - Normal Hepatic Function | Risdiplam M1 Metabolite - Mild Hepatic Impairment | Risdiplam M1 Metabolite - Normal Hepatic Function
Number analyzed (Participants) | 8 | 8 | 8 | 8
ng/mL | 21.7 (23.5) | 22.8 (46.9) | 3.73 (30.4) | 3.92 (36.3)
Statistical Analysis 1: Comparison: Risdiplam - Mild Hepatic Impairment vs Risdiplam - Normal Hepatic Function; Test type: Other — Descriptive statistics; Ratio of Geometric Least Squares Means = 0.950, 90% CI 2-sided [0.695 to 1.30]
Statistical Analysis 2: Comparison: Risdiplam M1 Metabolite - Mild Hepatic Impairment vs Risdiplam M1 Metabolite - Normal Hepatic Function; Test type: Other — Descriptive statistics; Ratio of Geometric Least Squares Means = 0.953, 90% CI 2-sided [0.715 to 1.27]

4. Primary Outcome: Part 2: AUCinf of Risdiplam and M1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- Risdiplam - Moderate Hepatic Impairment; Risdiplam M1 Metabolite - Moderate Hepatic Impairment: Participants with moderate hepatic impairment received a single dose of 5 mg risdiplam orally as a drinking solution on Day 1 after an overnight fast of at least 8 hours.
Arm/Group | Risdiplam - Moderate Hepatic Impairment | Risdiplam - Normal Hepatic Function | Risdiplam M1 Metabolite - Moderate Hepatic Impairment | Risdiplam M1 Metabolite - Normal Hepatic Function
Number analyzed (Participants) | 8 | 8 | 8 | 8
h*ng/mL | 1040 (29.2) | 971 (30.8) | 261 (23.4) | 275 (33.1)
Statistical Analysis 1: Comparison: Risdiplam - Moderate Hepatic Impairment vs Risdiplam - Normal Hepatic Function; Test type: Other — Descriptive statistics; Ratio of Geometric Least Squares Means = 1.08, 90% CI 2-sided [0.830 to 1.39]
Statistical Analysis 2: Comparison: Risdiplam M1 Metabolite - Moderate Hepatic Impairment vs Risdiplam M1 Metabolite - Normal Hepatic Function; Test type: Other — Descriptive statistics; Ratio of Geometric Least Squares Means = 0.947, 90% CI 2-sided [0.740 to 1.21]

5. Primary Outcome: Part 2: AUClast of Risdiplam and M1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Risdiplam - Moderate Hepatic Impairment | Risdiplam - Normal Hepatic Function | Risdiplam M1 Metabolite - Moderate Hepatic Impairment | Risdiplam M1 Metabolite - Normal Hepatic Function
Number analyzed (Participants) | 8 | 8 | 8 | 8
h*ng/mL | 1020 (29.7) | 947 (31.2) | 243 (24.9) | 259 (33.9)

6. Primary Outcome: Part 2: Cmax of Risdiplam and M1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Risdiplam - Moderate Hepatic Impairment | Risdiplam - Normal Hepatic Function | Risdiplam M1 Metabolite - Moderate Hepatic Impairment | Risdiplam M1 Metabolite - Normal Hepatic Function
Number analyzed (Participants) | 8 | 8 | 8 | 8
ng/mL | 29.9 (18.8) | 25.0 (30.2) | 4.10 (24.0) | 4.13 (22.5)
Statistical Analysis 1: Comparison: Risdiplam - Moderate Hepatic Impairment vs Risdiplam - Normal Hepatic Function; Test type: Other — Descriptive statistics; Ratio of Geometric Least Squares Means = 1.20, 90% CI 2-sided [0.962 to 1.49]
Statistical Analysis 2: Comparison: Risdiplam M1 Metabolite - Moderate Hepatic Impairment vs Risdiplam M1 Metabolite - Normal Hepatic Function; Test type: Other — Descriptive statistics; Ratio of Geometric Least Squares Means = 0.991, 90% CI 2-sided [0.810 to 1.21]

7. Secondary Outcome: Part 1: Time of the Maximum Observed Plasma Concentration (Tmax) of Risdiplam and M1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Risdiplam - Mild Hepatic Impairment | Risdiplam - Normal Hepatic Function | Risdiplam M1 Metabolite - Mild Hepatic Impairment | Risdiplam M1 Metabolite - Normal Hepatic Function
Number analyzed (Participants) | 8 | 8 | 8 | 8
hours (h) | 4.00 [2.00 to 4.00] | 4.00 [2.00 to 4.00] | 10.00 [4.00 to 24.00] | 10.00 [4.00 to 24.00]

8. Secondary Outcome: Part 1: Apparent Plasma Terminal Elimination Half-Life (t1/2) of Risdiplam and M1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Risdiplam - Mild Hepatic Impairment | Risdiplam - Normal Hepatic Function | Risdiplam M1 Metabolite - Mild Hepatic Impairment | Risdiplam M1 Metabolite - Normal Hepatic Function
Number analyzed (Participants) | 8 | 8 | 7 | 8
h | 41.3 (29.1) | 55.0 (16.2) | 32.9 (19.1) | 38.2 (18.7)

9. Secondary Outcome: Part 1: Percentage of Area Under the Plasma Concentration-Time Curve Due to Extrapolation (%AUCextrap) of Risdiplam and M1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage (%) of AUCextrap
Arm/Group | Risdiplam - Mild Hepatic Impairment | Risdiplam - Normal Hepatic Function | Risdiplam M1 Metabolite - Mild Hepatic Impairment | Risdiplam M1 Metabolite - Normal Hepatic Function
Number analyzed (Participants) | 8 | 8 | 7 | 8
Percentage (%) of AUCextrap | 2.34 (29.1) | 2.53 (32.8) | 7.49 (54.0) | 6.28 (38.7)

10. Secondary Outcome: Part 1: Terminal Elimination Rate Constant (λz=Lambda-Z) of Risdiplam and M1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h-1
Arm/Group | Risdiplam - Mild Hepatic Impairment | Risdiplam - Normal Hepatic Function | Risdiplam M1 Metabolite - Mild Hepatic Impairment | Risdiplam M1 Metabolite - Normal Hepatic Function
Number analyzed (Participants) | 8 | 8 | 7 | 8
h-1 | 0.0168 (29.1) | 0.0126 (16.2) | 0.0211 (19.1) | 0.0182 (18.7)

11. Secondary Outcome: Part 1: Apparent Total Clearance (CL/F) of Risdiplam
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Risdiplam - Mild Hepatic Impairment | Risdiplam - Normal Hepatic Function
Number analyzed (Participants) | 8 | 8
L/h | 6.31 (20.0) | 5.07 (35.2)

12. Secondary Outcome: Part 1: Molecular Weight-Adjusted Metabolite-to-Parent Ratio for AUCinf of Risdiplam M1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Risdiplam M1 Metabolite - Mild Hepatic Impairment | Risdiplam M1 Metabolite - Normal Hepatic Function
Number analyzed (Participants) | 7 | 8
Ratio | 0.258 (22.7) | 0.255 (12.0)

13. Secondary Outcome: Part 1: Molecular Weight-Adjusted Metabolite-to-Parent Ratio for Cmax of Risdiplam M1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Risdiplam M1 Metabolite - Mild Hepatic Impairment | Risdiplam M1 Metabolite - Normal Hepatic Function
Number analyzed (Participants) | 8 | 8
Ratio | 0.165 (29.4) | 0.164 (15.5)

14. Secondary Outcome: Part 1: Molecular Weight-Adjusted Metabolite-to-Parent Ratio for AUClast of Risdiplam M1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Risdiplam M1 Metabolite - Mild Hepatic Impairment | Risdiplam M1 Metabolite - Normal Hepatic Function
Number analyzed (Participants) | 8 | 8
Ratio | 0.244 (24.8) | 0.245 (13.8)

15. Secondary Outcome: Part 2: Tmax of Risdiplam and M1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Risdiplam - Moderate Hepatic Impairment | Risdiplam - Normal Hepatic Function | Risdiplam M1 Metabolite - Moderate Hepatic Impairment | Risdiplam M1 Metabolite - Normal Hepatic Function
Number analyzed (Participants) | 8 | 8 | 8 | 8
hours (h) | 2.00 [1.00 to 4.00] | 4.00 [1.00 to 4.00] | 24.00 [10.00 to 24.03] | 11.00 [4.00 to 24.00]

16. Secondary Outcome: Part 2: t1/2 of Risdiplam and M1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Risdiplam - Moderate Hepatic Impairment | Risdiplam - Normal Hepatic Function | Risdiplam M1 Metabolite - Moderate Hepatic Impairment | Risdiplam M1 Metabolite - Normal Hepatic Function
Number analyzed (Participants) | 8 | 8 | 8 | 8
h | 45.6 (28.0) | 49.9 (28.1) | 34.5 (24.3) | 35.0 (21.6)

17. Secondary Outcome: Part 2: %AUCextrap of Risdiplam and M1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage (%) of AUCextrap
Arm/Group | Risdiplam - Moderate Hepatic Impairment | Risdiplam - Normal Hepatic Function | Risdiplam M1 Metabolite - Moderate Hepatic Impairment | Risdiplam M1 Metabolite - Normal Hepatic Function
Number analyzed (Participants) | 8 | 8 | 8 | 8
Percentage (%) of AUCextrap | 1.90 (33.5) | 2.41 (30.5) | 6.58 (28.8) | 5.68 (23.6)

18. Secondary Outcome: Part 2: λz of Risdiplam and M1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h-1
Groups:
- Risdiplam - Moderate Hepatic Impairment: Participants with mild hepatic impairment received a single dose of 5 mg risdiplam orally as a drinking solution on Day 1 after an overnight fast of at least 8 hours.
Arm/Group | Risdiplam - Moderate Hepatic Impairment | Risdiplam - Normal Hepatic Function | Risdiplam M1 Metabolite - Moderate Hepatic Impairment | Risdiplam M1 Metabolite - Normal Hepatic Function
Number analyzed (Participants) | 8 | 8 | 8 | 8
h-1 | 0.0152 (28.0) | 0.0139 (28.1) | 0.0201 (24.3) | 0.0198 (21.6)

19. Secondary Outcome: Part 2: CL/F of Risdiplam and M1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Risdiplam - Moderate Hepatic Impairment | Risdiplam - Normal Hepatic Function
Number analyzed (Participants) | 8 | 8
L/h | 4.79 (29.2) | 5.15 (30.8)

20. Secondary Outcome: Part 2: Molecular Weight-Adjusted Metabolite-to-Parent Ratio for AUCinf of Risdiplam M1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Risdiplam M1 Metabolite - Moderate Hepatic Impairment | Risdiplam M1 Metabolite - Normal Hepatic Function
Number analyzed (Participants) | 8 | 8
Ratio | 0.239 (16.8) | 0.271 (10.3)

21. Secondary Outcome: Part 2: Molecular Weight-Adjusted Metabolite-to-Parent Ratio for Cmax of Risdiplam M1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Risdiplam M1 Metabolite - Moderate Hepatic Impairment | Risdiplam M1 Metabolite - Normal Hepatic Function
Number analyzed (Participants) | 8 | 8
Ratio | 0.131 (16.3) | 0.158 (15.0)

22. Secondary Outcome: Part 2: Molecular Weight-Adjusted Metabolite-to-Parent Ratio for AUClast of Risdiplam M1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Risdiplam M1 Metabolite - Moderate Hepatic Impairment | Risdiplam M1 Metabolite - Normal Hepatic Function
Number analyzed (Participants) | 8 | 8
Ratio | 0.227 (16.8) | 0.262 (10.0)

23. Secondary Outcome: Part 1 and Part 2: Percentage of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Up to 31 Days
Population: The safety population included all participants who received a dose of risdiplam.
Measure: Number; unit: Percentage of Participants
Groups:
- Part 1: Participants with mild hepatic impairment received a single dose of 5 mg risdiplam orally as a drinking solution on Day 1 after an overnight fast of at least 8 hours.
- Part 2: Participants with moderate hepatic impairment received a single dose of 5 mg risdiplam orally as a drinking solution on Day 1 after an overnight fast of at least 8 hours.
- Normal Hepatic Function Participants: Participants with normal hepatic function received a single dose of 5 mg risdiplam orally as a drinking solution on Day 1 after an overnight fast of at least 8 hours.
Arm/Group | Part 1 | Part 2 | Normal Hepatic Function Participants
Number analyzed (Participants) | 8 | 8 | 10
Percentage of Participants
  With at least one AE | 62.5 | 12.5 | 0.0
  With at least one SAE | 0.0 | 12.5 | 0.0

ADVERSE EVENTS:
Time Frame: Up to 31 days post-dose
Description: The safety population included all participants who received a dose of risdiplam.
Arm/Group | Mild Hepatic Impairment | Moderate Hepatic Impairment | Normal Hepatic Function
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/8 | 1/8 | 0/10
Other Adverse Events (participants affected / at risk) | 5/8 | 0/8 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mild Hepatic Impairment (N=8) | Moderate Hepatic Impairment (N=8) | Normal Hepatic Function (N=10)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mild Hepatic Impairment (N=8) | Moderate Hepatic Impairment (N=8) | Normal Hepatic Function (N=10)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights

DOCUMENTS (2):
  • Study Protocol (2019-01-08): https://cdn.clinicaltrials.gov/large-docs/65/NCT03920865/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-22): https://cdn.clinicaltrials.gov/large-docs/65/NCT03920865/SAP_001.pdf